CLINICAL TRIAL: NCT01214772
Title: the Effect of Unfractionated Heparin in Treatment of IVF-ET Failure
Brief Title: The Effect of Heparin in Treatment IVF-ET Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yazd Medical University (Other)
Collaborators: Yazd Research & Clinical Center for Infertility (Other)
Responsible Party: Dr Mehri Mashayekhy, Yazd Research and Clinical centre for infertility
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1378
Record Dates: First submitted 2010-09-28; First posted 2010-10-05 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-10

CONDITIONS: Pregnancy; Thrombophilia
Keywords: pregnancy; heparin; fertilization
MeSH Terms: conditions — Thrombophilia | interventions — Heparin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- heparin,pregnancy,IVF failure (Experimental): Women in the heparin arm are administered 5000 IU twice a day on the day of embryo transfer
  Interventions: Drug: heparin

INTERVENTIONS:
Drug: heparin — 5000 IU subcutaneously in the day of embryo transfer until 6 week after delivery

SUMMARY:
Embryo transfer failure is defined as ≥3 IVF-embryo transfer failures without pregnancy . In spite of transfer of 3 good quality embryos , just 20-30% of women undergoing IVF will achieve ongoing pregnancy . There are multiple factors that influence IVF-failure.

Autoantibodies may be one of the possible causes of IVF-failure , especially in unexplained and mechanical infertility .

In some studies , antiphospholipid antibody is considered as causative factor on implantation and embryo failure. However some investigators showed that combination therapy with heparin/aspirin in women with positive antiphospholipid antibody is not effective in improving of IVF-outcome . In prospective studies were not confirmed association between antiphospholipid antibody abnormalities and IVF-failure.

Recently has been relationship between thrombophilia and IVF and implantation failure.

The effect of unfractionated heparin in assisted reproductive technology (ART) cycles is prevention of thrombosis in implantation site . Although its effect is not restricted to anticoagulation and also can modulate apposition , adhesion , and penetration of embryo . Other advantages are decreasing thrombophilic risk in COH ( controlled ovarian hyperstimulation) cycles with administration of gonadotrophins . So heparin make better pregnancy rate in repeated IVF-ET failures.

There are few studies in regard to heparin effects on IVF cycles outcome . The purpose of this study is evaluation of unfractionated heparin effects on improvement of ART outcome .

This study was a prospective randomized controlled trial to assess whether administration of heparin would increased pregnancy rates in women with repeated ET-IVF failures.

DETAILED DESCRIPTION:
Introduction Embryo transfer failure is defined as ≥3 IVF-embryo transfer failures without pregnancy . In spite of transfer of 3 good quality embryos , just 20-30% of women undergoing IVF will achieve ongoing pregnancy . There are multiple factors that influence IVF-failure.

Autoantibodies may be one of the possible causes of IVF-failure , especially in unexplained and mechanical infertility .

In some studies , antiphospholipid antibody is considered as causative factor on implantation and embryo failure. However some investigators showed that combination therapy with heparin/aspirin in women with positive antiphospholipid antibody is not effective in improving of IVF-outcome . In prospective studies were not confirmed association between antiphospholipid antibody abnormalities and IVF-failure.

Recently has been relationship between thrombophilia and IVF and implantation failure.

The effect of unfractionated heparin in assisted reproductive technology (ART) cycles is prevention of thrombosis in implantation site . Although its effect is not restricted to anticoagulation and also can modulate apposition , adhesion , and penetration of embryo . Other advantages are decreasing thrombophilic risk in COH ( controlled ovarian hyperstimulation) cycles with administration of gonadotrophins . So heparin make better pregnancy rate in repeated IVF-ET failures There are few studies in regard to heparin effects on IVF cycles outcome . The purpose of this study is evaluation of unfractionated heparin effects on improvement of ART outcome .

Materials & Methods This study was a prospective randomized controlled trial to assess whether administration of unfractionated heparin would increased implantation and pregnancy rates in women with repeated ET-IVF failures or not . The study was performed at a reproduction center affiliated to a medical university. A total 86 patients who were candidate for IVF/ICSI with a history of three or more pervious IVF-ET failures enrolled in this study . The study was approved by the ethics committee of Research and Clinical Center for Infertility affiliated to Yazd Medical University of Medical Sciences . All patients were required to sign a written consent after the provision of complete information to them .

Treatment protocol All of the patients were treated with long protocol for ovarian stimulation. For pituitary suppression down regulation , the patients were treated with daily administration of 0.5 mg buserelin subcutaneous from day 21 of previous menstrual cycle. When desensitization was occurred, as evidenced by plasma E2 levels of ≤ 50 pg/ml and the absence of ovarian cyst on transvaginal ultrasound examination , buserelin was reduced to 0.25 mg/day and continued until the day of hCG administration. The COH was initiated with recombinant FSH or HMG 150 IU/day on the day 2 of menstrual cycle. Ovarian response was monitored by serial ultrasound examinations and evaluation of serum E2 levels, and then gonadotropin doses adjustment was done as required. Urinary HCG 10000 IU was administered when ≥3 follicles more than 18 mm.

Oocyte retrieval was performed 34-36 hours after hCG injection and IVF or ICSI was performed.

one to three top-quality embryos were transferred 48 hours after oocyte retrieval under ultrasound guidance , with a CCD embryo transfer catheter. At the same time , patients (n=86) were randomized to two groups using a computer-generated randomization . Group A ( n=43) included the patients who received unfractionated heparin 5000 IU twice a day subcutaneous injection . Treatment was started from the day of embryo transfer until 14 days after ET . If β-hCG was positive , the unfractionated heparin was continued until 6 weeks postpartum . Group B ( n=43 ) did not receive any antithrombotic drugs.

Luteal phase support was started with administration of progesterone 100 mg daily intramuscular on the day of oocyte retrieval in two groups and continued until the documentation of fetal heart activity on ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were 19-35 years old
* basal FSH < 10 IU/l
* body mass index ( BMI ) < 29 Kg/m²
* presence of both ovaries
* three or more pervious IVF-ET failures
* Top-quality embryos for transfer .

Exclusion Criteria:

* Women with polycystic ovary syndrome ( PCOS)
* endometriosis
* hydrosalpinx
* chronic systemic disease( liver, renal , thyroid and thrombocytopenia ) ●Abnormal uterine cavity
* sever male factor ( azospermia )
* Patients who had contraindication for unfractionated heparin therapy .

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
chemical pregnancy rate | until 12th gestational week

SECONDARY OUTCOMES:
clinical pregnancy rate | until 12 gastational week

CONTACTS AND LOCATIONS:
Overall Officials: Mehri Mashayekhy, infertility fellowship, Principal Investigator — Yazd Research and Clinical Centre for Infertility
Locations (1):
- Yazd Research and Clinical Centre for Infertility, Yazd, Yazd Province, Iran